CLINICAL TRIAL: NCT04087070
Title: Blood Pressure Estimation Using Noninvasive Biosignals During Pediatric Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Other Study IDs: H-1907-088-1049
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Blood Pressure; Pediatrics; Electrocardiography; Accelerometer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- biosignal derived blood pressure: Blood pressure is measured by an automated oscillometric device or arterial waveform from IntelliVue MX800 Bedside patient monitor (Philips Healthcare, Amsterdam, Netherlands).
  Following parameters will be measured by non-invasive electrocardiogram (ECG), photoplethysmograph (PPG), and an accelerometer on the chest and will be used to estimate the biosignal derived blood pressure.
  1. PAT(time between R peak of ECG and beginning of the pulse of PPG)
  2. PEP(time between R peak of ECG and peak of accelerometer signal)
  3. PTT(PAT-PEP)
  Interventions: Device: Biosignal measurements

INTERVENTIONS:
Device: Biosignal measurements — Following parameters will be measured by non-invasive electrocardiogram (ECG), photoplethysmograph (PPG), and an accelerometer on the chest and will be used to estimate the biosignal derived blood pressure.
  1. PAT(time between R peak of ECG and beginning of the pulse of PPG)
  2. PEP(time between R peak of ECG and peak of accelerometer signal)
  3. PTT(PAT-PEP)

SUMMARY:
The aim of this study is to estimate blood pressure in pediatric patients using a non-invasive electrocardiogram (ECG), photoplethysmograph (PPG), and an accelerometer on the chest.

DETAILED DESCRIPTION:
Blood pressure is measured by an automated oscillometric device or arterial waveform from IntelliVue MX800 Bedside patient monitor (Philips Healthcare, Amsterdam, Netherlands).

Following parameters will be measured by non-invasive electrocardiogram (ECG), photoplethysmograph (PPG), and an accelerometer on the chest and will be used to estimate the biosignal derived blood pressure.

1. PAT(time between R peak of ECG and beginning of the pulse of PPG)
2. PEP(time between R peak of ECG and peak of accelerometer signal)
3. PTT(PAT-PEP)

The algorithm of the biosignal derived blood pressure will be made using the MATLAB 2016b(Mathworks, Natick, MA) program.

The agreement between the non-invasive blood pressure and the biosignal derived blood pressure will be analyzed using Cohen's Kappa or Bland-Altman plot.

ELIGIBILITY:
Inclusion Criteria:

* ASA(American Society of Anesthesiologist) Class I, II
* Scheduled for elective surgery under general anesthesia

Exclusion Criteria:

* History of cardiovascular disease
* History of thoracic cavity disease
* Unable to measure blood pressure

Max Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: ASA class I, and II pediatric patients (<12 years) scheduled for elective surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-28 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Systolic and diastolic Blood pressure | During general anesthesia, up to 12 hours
  Systolic and diastolic blood pressure by automated oscillometric device or arterial waveform from IntelliVue MX800 Bedside patient monitor (Philips Healthcare, Amsterdam, Netherlands).

SECONDARY OUTCOMES:
Electrocardiogram wave | During general anesthesia, up to 12 hours
  Electrocardiogram wave
photoplethysmograph wave | During general anesthesia, up to 12 hours
  photoplethysmograph wave
accelerometer signal | During general anesthesia, up to 12 hours
  accelerometer signal

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, MD.PhD, Principal Investigator — Department of Anesthesiology and Pain Medicine, Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
We art not planning to share individual participant data available to other researchers

REFERENCES:
- [Background] Yoon Y, Cho JH, Yoon G. Non-constrained blood pressure monitoring using ECG and PPG for personal healthcare. J Med Syst. 2009 Aug;33(4):261-6. doi: 10.1007/s10916-008-9186-0. PMID 19697692